CLINICAL TRIAL: NCT04748263
Title: Eye Gaze Strategies During Facial Emotion Recognition in Neurodegenerative Diseases: Links With Neuropsychiatric Disorders (EYE-ToM Study)
Acronym: EYE-ToM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Princesse Grace (Other)
Collaborators: Association de Recherche Bibliographique pour les Neurosciences (Other)
Responsible Party: Sponsor
Other Study IDs: 15-05
Record Dates: First submitted 2021-01-26; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer's Dementia; Parkinson Disease(PD); Fronto-Temporal Dementia
Keywords: Eye-Tracking; Neuropsychological evaluations
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Fronto-Temporal Dementia (FTD): 10 subjects Standard neuropsychological evaluations. Standard Eye-Tracking paradigms.
  Interventions: Other: No intervention. Only survey and normal use of eye-tracking
- Alzheimer's Dementia (AD): 20 subjects Standard neuropsychological evaluations. Standard Eye-Tracking paradigms.
  Interventions: Other: No intervention. Only survey and normal use of eye-tracking
- Parkinson's Disease (PD): 20 subjects Standard neuropsychological evaluations. Standard Eye-Tracking paradigms.
  Interventions: Other: No intervention. Only survey and normal use of eye-tracking
- Healthy volunteers: 20 subjects Standard neuropsychological evaluations. Standard Eye-Tracking paradigms.
  Interventions: Other: No intervention. Only survey and normal use of eye-tracking

INTERVENTIONS:
Other: No intervention. Only survey and normal use of eye-tracking — The study is conducted in accordance with usual practices of eye-tracking and neuropsychological evaluations carried out at the Center Rainier III.
  Eye-Tracker® is used at the Centre Rainier III since August 2014. It is a non-invasive device for eye movements recording, allowing doctors and researchers to measure standard parameters related to eye movements. Developed by the Eye Brain Company (France), this is a Class IIa medical device, CE marking, according to Annexe IX of the directive 93/42/CE.

SUMMARY:
It is commonly admitted that social cognition impairment, like deficit in facial emotion recognition or misinterpretation of others' intentions (Theory of Mind), are associated with social behavior disorders.

This kind of disorders are observed in Fronto-Temporal Dementia (FTD), Alzheimer's Dementia (AD) and Parkinson's Disease (PD), with severe deficits in FTD and lighter deficits in AD and PD.

One explanation might be that patients apply inappropriate visual exploration strategies to decode emotions and intentions of others.

This study aims to test this hypothesis and further to analyse whether different patterns emerge from these pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized or coming to perform a consultation, for whom an Eye-Tracking examination is indicated as part of routine care.
* Sufficient written and oral expression in French.
* Written informed consent signed by the patient.
* For the control group: No cognitive impairment (non pathological MMSE (according to age, gender and socio-cultural level), no neurological history, and no psychiatric history (especially anxiety and depressive disorders).
* For the FTD group: Patient diagnosed according to revised Rascovsky et al. 2011., no neurological history (excepted diagnosed FTD), and no psychiatric history (excepted those related to diagnosed FTD).
* For the AD group: Patient diagnosed according to DSM-IV-TR criteria, no neurological history (excepted diagnosed AD), and no psychiatric history (excepted those related to diagnosed AD).
* For the PD group: Patient diagnosed according to NINDS criteria, no neurological history (excepted diagnosed PD), and no psychiatric history (excepted those related to diagnosed PD).

Exclusion Criteria:

* General anaesthesia within 3 months.
* Ophthalmological problems preventing a video-oculography examination.
* Oculomotor disorders such as "fixation disorders" or "ocular tracking disorders".
* Cognitive disorders of the type: visual agnosia, visuo-spatial disorder, visuo-perceptual disorder or aphasia.
* History of stroke.
* History of alcohol or drug abuse.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient 45 years old and above healthy or with FTD, AD or PD pathology
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Eye gaze strategies (number of eye fixation) during Affective Theory of Mind (ToM) | Baseline
  Comparison of gaze patterns between control group and pathological groups, during Affective ToM task Evaluation criteria: number of eye fixation. Eye movements were recorded with an eye-tracking device. Affective ToM was assessed using the " Reading the Mind in the Eyes " test (Baron-Cohen 2001).
Eye gaze strategies (duration of eye fixations) during Affective Theory of Mind (ToM) | Baseline
  Comparison of gaze patterns between control group and pathological groups, during Affective ToM task.
  Evaluation criteria: duration of eye fixations. Eye movements were recorded with an eye-tracking device. Affective ToM was assessed using the " Reading the Mind in the Eyes " test (Baron-Cohen 2001).
Eye gaze strategies (response times) during Affective Theory of Mind (ToM) | Baseline
  Evaluation criteria: time to answer for each picture (in second). It was recorded using the eye-tracking device.
  Affective ToM was assessed using 36 pictures from the " Reading the Mind in the Eyes " test (Baron-Cohen 2001), with a maximum of 8 seconds of response time per picture.
Eye gaze strategies (number of eye fixation) during Facial emotion recognition (FER) | Baseline
  Comparison of gaze patterns between control group and pathological groups, during Facial emotion recognition tasks.
  Evaluation criteria: number of eye fixation. Eye movements were recorded with an eye-tracking device. FER was assessed using some pictures from the Ekman Faces task (1976).
Eye gaze strategies (duration of eye fixation) during Facial emotion recognition (FER) | Baseline
  Comparison of gaze patterns between control group and pathological groups, during Facial emotion recognition tasks.
  Evaluation criteria: duration of eye fixations. Eye movements were recorded with an eye-tracking device. FER was assessed using some pictures from the Ekman Faces task (1976).
Eye gaze strategies (response times) during Facial emotion recognition (FER) | Baseline
  Comparison of gaze patterns between control group and pathological groups, during Facial emotion recognition tasks.
  Evaluation criteria: time to answer for each picture (in second). It was recorded using the eye-tracking device.
  Facial emotion recognition was assessed using 28 pictures from The Ekman Faces task (1976), with a maximum of 8 seconds of response time per picture.

SECONDARY OUTCOMES:
Facial emotion recognition (FER) performances | Baseline
  Affective ToM performances, and behavioral disorders. Evaluation criteria: Scores (/28) and sub-score (/6) to Ekman Faces task (1976).
  The Ekman Faces task (1976) tests the recognition of the six facial basic emotions and neutral faces. There were four pictures per emotion, for a total of 28. For each picture, participants were asked to select one of the seven labels (anger, disgust, fear, sadness, happiness, surprise and neutral)
Affective ToM performances | Baseline
  To study correlations between eye gaze strategies, Facial emotion recognition and Affective ToM performances, and behavioral disorders.
  Evaluation criteria: Scores to the " Reading the Mind in the Eyes " test (Baron-Cohen 2001). 36 black-and-white photographs of the eye area of faces. Subjects are asked to choose which word, among four options, best described what the character in the photograph was thinking or feeling. For this task, four scores were obtained: a total score (/36) and three emotional valence sub-scores: positive (/8), neutral (/16) and negative (/12).
Behavioral disorders. | Baseline
  To study correlations between eye gaze strategies, Facial emotion recognition and Affective ToM performances, and behavioral disorders.
  Evaluation criteria: Neuropsychiatric Inventory (NPI), a scale that includes ten behavioral items (delusions, hallucinations, agitation, depression, anxiety, euphoria, apathy, disinhibition, irritability and aberrant motor behaviors) and two neurovegetative symptoms (sleep and appetite disorders). Both the frequency (/5) and the severity (/3) of each behavior were determined and a score was calculated by multiplying the frequency and the severity of each behavior observed during the last month.

CONTACTS AND LOCATIONS:
Overall Officials: Alain PESCE, MD-PHD, Principal Investigator — CH Princesse Grace; Sandrine LOUCHART de la CHAPELLE, MD, Principal Investigator — CH Princesse Grace

IPD SHARING:
Plan to Share IPD: No